CLINICAL TRIAL: NCT03705455
Title: Immunization Schedule Alert Platform: Determining ISAP SMS Efficacy in Improving Childhood Immunization Timeliness and Completeness in Nigeria
Brief Title: Immunization Schedule Alert Platform
Acronym: ISAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lifespan Healthcare Resource Limited (Other)
Responsible Party: Principal Investigator, Dr.Ihedioha Emmanuel Chukwunwike, Principal Investigator, Lifespan Healthcare Resource Limited
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPP1182651
Record Dates: First submitted 2018-10-09; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Immunization

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ISAP SMS (Active Comparator): ISAP SMS will be sent to enrolled caregivers
  Interventions: Behavioral: ISAP SMS
- No ISAP SMS (No Intervention): No ISAP SMS will be sent to enrolled caregivers

INTERVENTIONS:
Behavioral: ISAP SMS — ISAP SMS is a text message for caregivers use that provides immunization schedule and vaccine availability at the nearest immunization clinic.
  Arms: ISAP SMS

SUMMARY:
The ISAP study is investigating the efficacy of SMS messages in improving routine childhood Immunization timeliness and completeness in Nigeria.

DETAILED DESCRIPTION:
The ISAP - Immunization Schedule Alert Platform study is investigating the efficacy of ISAP SMS exposure to Caregivers with children( who have fulfilled our inclusion criteria) due for routine childhood Immunisation in influencing decision for timely and complete Immunization uptake. ISAP SMS messages contains information on the Immunization appointment schedule, time ,vaccine to be administered and the address of the Immunization centre.

ELIGIBILITY:
Inclusion Criteria:

Caregiver with child due for birth dose vaccination or at 6weeks-OPV1,Penta1,PCV1,Rota1.

Exclusion Criteria: Caregiver with child who have already had OPV1,Penta1,PCV1and Rota1.

-

Ages: 6 Weeks to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1800 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of timely and complete vaccine uptake after ISAP SMS Intervention | 12 months
  Proportion of timely and complete vaccine uptake after ISAP SMS Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Ihedioha, MBBS, Principal Investigator — Lifespan Healthcare Resource
Locations (1):
- Nkanu East Health centre Immunization clinic, Enugu, Nigeria

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276